CLINICAL TRIAL: NCT02810834
Title: Understanding the Impact of School-Based Physical Activity Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: R01HD080180 (NIH); 1R01HD080180-01A1 (NIH)
Record Dates: First submitted 2015-05-11; First posted 2016-06-23 (Estimated); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Physical Activity
Keywords: Executive Function; Academic Performance
MeSH Terms: conditions — Motor Activity | interventions — Walking

ARMS (3):
- Walking/Running Program (Experimental): Walking/running/jogging program; school-based.
  Interventions: Behavioral: Walking/Running program
- Classroom activity break program (Experimental): Classroom physical activity break program; school-based.
  Interventions: Behavioral: Classroom physical activity break program
- Control (No Intervention): Control/Delayed Intervention

INTERVENTIONS:
Behavioral: Walking/Running program — Participants will receive a behavioral intervention that consists of a school-based, walking/running/jogging program. Participants work to accumulate miles towards a goal of at least 100 miles, over the course of the school year. Program will be implemented through a "champion" in the school and structured/scheduled according to the schools resources (before, during, or after school). Miles are tracked at the school level, and incentives are provided for participants' completion of set milestones (25, 50, 75, and 100 miles).
  The intervention will run over two school years (approximately 16 months)
  Other Names: 100 Mile Club
  Arms: Walking/Running Program
Behavioral: Classroom physical activity break program — Participants will receive a behavioral intervention that consists of a classroom-based, physical activity break program. Classroom teachers, paraprofessionals, and other school staff will lead short (5-15 minute) activity breaks that include both higher intensity (ex. jumping jacks, squats) and low-intensity (ex. stretching, yoga) activities. Classrooms will be encouraged to integrate at least one short break per day. Activities are connected to national Common Core academic standards so that breaks can be integrated with academics.
  The intervention will run over two school years (approximately 16 months)
  Other Names: Just Move
  Arms: Classroom activity break program

SUMMARY:
The central hypothesis of the Fueling Learning Through Exercise (FLEX) study is two innovative school-based physical activity programs (a walking/running program and a classroom activity break program) will increase school-time and total daily minutes children engage in moderate-to-vigorous physical activity, relative to controls, and that children who attend schools with these PA programs will demonstrate improved cognitive functioning, academic achievement, and attendance, relative to controls.

DETAILED DESCRIPTION:
The FLEX Study is a three-year, randomized control trial that seeks to understand how two different innovative school-based physical activity (PA) programs influence not only children's time spent in MVPA but also their cognitive and academic outcomes. The FLEX Study will be implemented and evaluated by researchers from Tufts University. The project is funded by the National Institutes of Health.

Schools participating in the study will be randomly assigned to receive a walking/running program, a classroom physical activity program, or no program (control) during first year and a half of the study. Third and fourth grade children will be enrolled in the study.

Physical activity will be assessed objectively using accelerometry. Additional measurements will include: BMI/BMI-z (measured height and weight), diet and physical activity questionnaires, cognitive functioning (tests of working memory and inhibitory control).

ELIGIBILITY:
Inclusion Criteria:

Children participants 3rd or 4th grade student in participating school (during first school year of study)

Exclusion Criteria:

Not a 3rd or 4th grade student

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1182 (Actual)
Dates: Start 2014-09; Primary Completion 2017-06-23 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
School-time and total daily MVPA | 5 months and 1.5 years
  Changes in minutes of school-time and total daily moderate-to-vigorous physical activity (MVPA) among third-fifth graders participating in innovative school-based physical activity programs, compared to controls

SECONDARY OUTCOMES:
Cognitive performance | 5 months and 1.5 years
  Changes in cognitive performance, as measured by standard tests of executive function, among third-fifth graders participating in innovative
Academic achievement | 5 months and 1.5 years
  Changes in academic achievement, as measured by standardized tests (English language art and math), among third-fifth graders participating in innovative

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer M Sacheck, PhD, Principal Investigator — Tufts University
Locations (1):
- Gerald J. and Dorothy R. Friedman School of Nutrition Science and Policy, Tufts University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Neil-Sztramko SE, Caldwell H, Dobbins M. School-based physical activity programs for promoting physical activity and fitness in children and adolescents aged 6 to 18. Cochrane Database Syst Rev. 2021 Sep 23;9(9):CD007651. doi: 10.1002/14651858.CD007651.pub3. PMID 34555181
- [Derived] Sacheck JM, Wright CM, Amin SA, Anzman-Frasca S, Chomitz VM, Chui KK, Duquesnay PJ, Nelson ME, Economos CD. The Fueling Learning Through Exercise Study Cluster RCT: Impact on Children's Moderate-to-Vigorous Physical Activity. Am J Prev Med. 2021 Jun;60(6):e239-e249. doi: 10.1016/j.amepre.2021.01.002. Epub 2021 Mar 26. PMID 33781620
- [Derived] Wright CM, Chomitz VR, Duquesnay PJ, Amin SA, Economos CD, Sacheck JM. The FLEX study school-based physical activity programs - measurement and evaluation of implementation. BMC Public Health. 2019 Jan 16;19(1):73. doi: 10.1186/s12889-018-6335-3. PMID 30651117
- [Derived] Amin SA, Duquesnay PJ, Wright CM, Chui K, Economos CD, Sacheck JM. The Association Between Perceived Athletic Competence and Physical Activity: Implications for Low-Income Schoolchildren. Pediatr Exerc Sci. 2018 Aug 1;30(3):433-440. doi: 10.1123/pes.2017-0242. Epub 2018 Mar 15. PMID 29543115
- [Derived] Wright CM, Duquesnay PJ, Anzman-Frasca S, Chomitz VR, Chui K, Economos CD, Langevin EG, Nelson ME, Sacheck JM. Study protocol: the Fueling Learning through Exercise (FLEX) study - a randomized controlled trial of the impact of school-based physical activity programs on children's physical activity, cognitive function, and academic achievement. BMC Public Health. 2016 Oct 13;16(1):1078. doi: 10.1186/s12889-016-3719-0. PMID 27737676